CLINICAL TRIAL: NCT05577286
Title: Therapeutic Effects of Plyometric Exercises in Children With Type 1 Diabetis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Assist Prof. Physical therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: type 1 diabetes
Record Dates: First submitted 2022-09-27; First posted 2022-10-13 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes mellitus; type 1 1 Diabetes mellitus; plyometric exercises; balance; muscle strength
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): 15 Children with type 1 Diabetes mellitus in this group will receive the regular medical treatment without change of their daily activity routine
  Interventions: Other: regular care
- plyometric group (Experimental): 15 Children with type 1 Diabetes mellitus in this group will receive the regular medical treatment as in control group in addition to a designed plyometric training program for 30 minutes, three times a week for two successive months.
  Interventions: Other: regular care; Other: plyometric training

INTERVENTIONS:
Other: regular care — the regular medical treatment without change of their daily activity routine
Other: plyometric training — designed plyometric training program for 30 minutes, three times a week for two successive months
  Arms: plyometric group

SUMMARY:
Despite the benefits of physical rehabilitation among adults and children with chronic illness such as Diabetes mellitus avoid engaging in different physical activities especially pediatric population. Most of the children with type 1 Diabetes mellitus receive their medical treatment and follow-up with no change of their functional performance.

DETAILED DESCRIPTION:
We still lack the evidence of plyometric exercises in pediatric population with Diabetes mellitus . Therefore, the primary aim of this study is to explore the effects of plyometric exercises on blood glucose level, balance and muscle strength in children with 1 Diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Age will range from six to 10 years
* Both sexes
* Chronicity of the disease ranges from 3 to <5 years.
* Controlled diabetes with insulin dosage described by physician.

Exclusion Criteria:

* Heriderty sensory or autonomic peripheral neuropathy.
* Unstable cardio-vascular disorders
* History of fractures or surgery in the lower extremities in the past 12 months.
* Diagnosed with other hormonal diseases.
* Children who practice regular sports.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
muscle strength | after 3 successive months
  assessment of hip, knee and ankle muscles by The Laffayette manual muscle testing (model 01163 USA) which measure strength in kG.
balance | after 3 successive months
  assessment of balance by The Human Assessment Computer (HUMAC), a computerized dynamic posturography (commuter sports medicine, Inc., Stoughton, MA).

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Mahmoud Sanad, Phd, Study Chair — Cairo university, faculty of physical therapy; Samya M Aly Hussein, B.Sc., Principal Investigator — Cairo university, faculty of physical therapy; Aboalnaga A Abdelrahim Hamed, Study Director — Cairo university, faculty of physical therapy